CLINICAL TRIAL: NCT03042832
Title: Testing the Leadership and Organizational Change for Implementation (LOCI) Intervention in Substance Abuse Treatment Programs
Brief Title: Testing the Leadership and Organizational Change for Implementation (LOCI) Intervention
Acronym: LOCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Gregory Aarons, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 141134
Record Dates: First submitted 2016-10-25; First posted 2017-02-03 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Substance Use Disorder; Mental Health Disorder
Keywords: Leadership; Organizational Climate; Implementation; Implementation Climate; Motivational Interviewing; Fidelity
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Intention To Treat (ITT) model with clinics randomized to LOCI vs Webinar control
Oversight: Data Monitoring Committee: No

ARMS (2):
- LOCI (Experimental): Leadership development with coaching and organizational change support
  Interventions: Behavioral: LOCI
- Internet Based Training (Active Comparator): Internet based Webinar leadership training
  Interventions: Behavioral: Internet Based Webinar Leadership Training

INTERVENTIONS:
Behavioral: LOCI — Leadership development with coaching and organizational change support
  Arms: LOCI
Behavioral: Internet Based Webinar Leadership Training — Internet Based Webinar Leadership Training
  Arms: Internet Based Training

SUMMARY:
This study will test the effects of the Leadership and Organizational Change for Implementation (LOCI) intervention in facilitating evidence-based practice (EBP) implementation in substance use disorder (SUD) and HIV services settings. LOCI improves implementation leadership and organizational support to develop strategic climate for EBP implementation. Greater efficiency and effectiveness of EBP implementation will improve the public health impact of evidence-based health and allied healthcare innovations and lead to greater effectiveness of SUD and HIV services.

Project Terms:

DETAILED DESCRIPTION:
Effective implementation of evidence-based practices (EBPs) to address complex and widespread public health issues, such as substance use disorders (SUDs) and HIV, remains a substantial challenge. Leadership and organizational context are associated with implementation climate and attitudes toward EBP, as well as clinical outcomes such as client satisfaction and quality of life. While there are many leadership development approaches, they are often not based on empirically supported approaches and curricula, nor are they specifically designed to develop strategic climates for EBP implementation. This project addresses these concerns and advances implementation science by testing the effects of the Leadership and Organizational Change for Implementation (LOCI) intervention. The goals of the LOCI intervention are to improve general leadership and implementation leadership and utilize organizational strategies to create a positive strategic organizational climate for EBP implementation. These should lead to more positive SUD treatment provider attitudes and behaviors that support EBP implementation outcomes of intervention fidelity and implementation process. Consistent with the Exploration, Preparation, Implementation, Sustainment (EPIS) conceptual framework, LOCI creates change at multiple levels within a provider organization (e.g., executives/mid- managers, workgroup leader, service provider) to foster a context supportive of EBP implementation and sustainment. Initial support for the feasibility, acceptability, and utility of the LOCI intervention have been successfully demonstrated in an NIH supported pilot study (R21MH082731, PI: Aarons). The proposed study will test whether LOCI can achieve change in outcomes of general and implementation leadership, implementation climate, implementation process, and EBP fidelity in SUD treatment agencies. Seventy-two workgroup leaders and their providers (i.e., subordinates) will be randomized to either the LOCI condition or a Webinar control condition. All direct SUD treatment providers in both conditions will receive training in Motivational Interviewing (MI), a leading EBP for SUD and HIV prevention and treatment. The test of LOCI will occur within four agencies that provide SUD treatment at multiple sites across California. The test of the LOCI intervention will include SUD service providers (n=320), workgroup leaders (n=60), and agency executives/mid-managers (n=16). Hypotheses will be tested comparing LOCI and control group outcomes of leadership, implementation climate, psychological safety climate, provider attitudes and behaviors, MI fidelity, and implementation process. The proposed study will provide a practical implementation strategy that can be utilized to improve workgroup leadership and strategic climate for EBP implementation.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder treatment service providers, supervisors, agency executives/managers
* Supervisors will be the only individuals eligible to participate in the experimental (LOCI) or control condition (internet based) leadership intervention.
* Only supervisors in the experimental (LOCI) condition will be eligible to participate in focus groups.
* Only agency executives/managers participating in the organizational strategy development meetings of the LOCI intervention condition will be eligible to participate in interviews.

Exclusion Criteria:

* Personnel not providing or supervising direct services (e.g., administrative staff) are not included as most of the measures will not be applicable to these staff.
* Participants must be at least 18 years of age and employed at one of the participating agencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Implementation Leadership | 12 months
  The Implementation Leadership Scale (ILS: Aarons et al., 2014) is a brief 12-item measure with four subscales: Proactive Leadership, Knowledgeable Leadership, Supportive Leadership, and Perseverant Leadership. This measure will be included in the survey for providers, workgroup supervisors, and managers/executives. Data will be aggregated at the workgroup level.
Full Range Leadership | 12 months
  The Multifactor Leadership Questionnaire (MLQ: Bass & Avolio, 1990) is one of the most widely used measures of leadership in organizations. The MLQ assesses transformational and transactional leadership. This measure will be included in the survey for providers, workgroup supervisors, and managers/executives.

SECONDARY OUTCOMES:
Implementation Climate | 12 months
  1. The Implementation Climate Scale (ICS; Ehrhart, Aarons, & Farahnak, 2015) will be used to assess organizational climate for implementation. ICS dimensions include 1) focus on EBP, 2) educational support for EBP, 3) recognition for EBP, 4) rewards for EBP, 5) selection for EBP, and 6) selection for openness. Data will be aggregated at the workgroup level.
Attitudes Toward Evidence-Based Practice | 12 months
  The Evidence-Based Practice Attitude Scale (EBPAS; Aarons 2004 will assess individuals attitudes toward EBP. The EBPAS is a 15-item measure with four subscales that assess attitudes toward adoption of EBP as a function of perceived appeal EBP, Requirements to use EBP, provider Openness, and perceived Divergence between EBP and usual care. The EBPAS is an individual level construct and will not be aggregated to the workgroup level.
Implementation Citizenship Behavior | 12 months
  The Implementation Citizenship Behavior Scale (ICBS; Ehrhart, Aarons, Farahnak, 2015) [69] will be used to assess individuals EBP implementation citizenship behavior. The ICBS was adapted from an existing reliable and valid measure of safety citizenship behavior in the workplace [76] and assesses the extent to which individual workgroup members go above and beyond minimum requirements to support successful EBP implementation in regard to helping others and keeping informed. The ICBS is an individual level construct and will not be aggregated to the workgroup level.
Fidelity | 12 months
  MI Coaching Rating Scale (MI-CRS; Naar-King & Suarez, 2011) will be used. This scale was developed based on the Motivational Interviewing Treatment Integrity Instrument (MITI) [78] that has demonstrated inter-rater reliability and differentiates between MI and usual care. Data will be aggregated at the workgroup level.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarons GA, Ehrhart MG, Moullin JC, Torres EM, Green AE. Testing the leadership and organizational change for implementation (LOCI) intervention in substance abuse treatment: a cluster randomized trial study protocol. Implement Sci. 2017 Mar 3;12(1):29. doi: 10.1186/s13012-017-0562-3. PMID 28253900
- [Derived] Aarons GA, Sklar M, Ehrhart MG, Roesch S, Moullin JC, Carandang K. Randomized trial of the leadership and organizational change for implementation (LOCI) strategy in substance use treatment clinics. J Subst Use Addict Treat. 2024 Oct;165:209437. doi: 10.1016/j.josat.2024.209437. Epub 2024 Jun 10. PMID 38866139